CLINICAL TRIAL: NCT03630887
Title: Prevention of Perioperative Hypothermia in Patients Submitted to Transurethral Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Negrin University Hospital (Other)
Collaborators: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Ángel Becerra, Principal Investigator, Dr. Negrin University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RTU-2018-153-1
Record Dates: First submitted 2018-08-08; First posted 2018-08-15 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Hypothermia; Anesthesia; Perioperative/Postoperative Complications; Complication of Anesthesia; Temperature Change, Body; Anaesthesia Complication; Transurethral Resection Syndrome
Keywords: Prewarming; Tympanic temperature; Transurethral Resection
MeSH Terms: conditions — Hypothermia; Postoperative Complications; Body Temperature Changes; Transurethral resection syndrome

STUDY DESIGN:
Intervention Model Description: We will compare different time periods: 0 minutes (control group), 15 minutes, 30 minutes and 45 minutes.
  Sample size was authorized by IRB to be changed from 144 to 244 (61 patients per group) due to possible missing data.
Who Masked: Care Provider, Investigator
Masking Description: Randomization will be carried out by a collaborator investigator using a computer program (Excel 2016) when a new patient is included into the clinical trial. This collaborator investigator will call by phone the nurse in charge of receiving the patient in the preanesthetic room, telling this nurse how long prewarming has to be given to the patient: 0 minutes (no prewarming), 15 minutes, 30 minutes or 45 minutes, according to the group given by the computer program. This collaborator investigator will not provide clinical care to the patient. Thus, principal investigator will not be able to know how long prewarming will be given by the nurse to the patient (chosen by the computer program and organized by a collaborator investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Non-active prewarming. Patients will be actively warmed during the intraoperative period. Tympanic thermometer (Genius 2 Tympanic Thermometer and Base, Covidien Ltd, Mansfield, USA) will be used to measure the temperature throughout the perioperative period.
- Prewarming during 15 minutes (Experimental): Active Prewarming will be performed during 15 minutes, using a forced-air blanket (WarmTouch lower body blanket, Covidien Ltd, Mansfield, USA) over the whole body and connected to a forced-air warmer (WarmTouch Model 5900, Covidien Ltd, Mansfield, USA). Patients will be actively warmed during the intraoperative period. Tympanic thermometer (Genius 2 Tympanic Thermometer and Base, Covidien Ltd, Mansfield, USA) will be used to measure the temperature throughout the perioperative period.
  Interventions: Device: WarmTouch Model 5900, Covidien Ltd, Mansfield, USA
- Prewarming during 30 minutes (Experimental): Active Prewarming will be performed during 30 minutes, using a forced-air blanket (WarmTouch lower body blanket, Covidien Ltd, Mansfield, USA) over the whole body and connected to a forced-air warmer (WarmTouch Model 5900, Covidien Ltd, Mansfield, USA). Patients will be actively warmed during the intraoperative period. Tympanic thermometer (Genius 2 Tympanic Thermometer and Base, Covidien Ltd, Mansfield, USA) will be used to measure the temperature throughout the perioperative period.
  Interventions: Device: WarmTouch Model 5900, Covidien Ltd, Mansfield, USA
- Prewarming during 45 minutes (Experimental): Active Prewarming will be performed during 45 minutes, using a forced-air blanket (WarmTouch lower body blanket, Covidien Ltd, Mansfield, USA) over the whole body and connected to a forced-air warmer (WarmTouch Model 5900, Covidien Ltd, Mansfield, USA). Patients will be actively warmed during the intraoperative period. Tympanic thermometer (Genius 2 Tympanic Thermometer and Base, Covidien Ltd, Mansfield, USA) will be used to measure the temperature throughout the perioperative period.
  Interventions: Device: WarmTouch Model 5900, Covidien Ltd, Mansfield, USA

INTERVENTIONS:
Device: WarmTouch Model 5900, Covidien Ltd, Mansfield, USA — Forced-air warming will be applied in the preanesthetic room during different time periods.
  Arms: Prewarming during 15 minutes; Prewarming during 30 minutes; Prewarming during 45 minutes

SUMMARY:
Hypothermia is a frequent perioperative complication. When the negative effects of anesthesia on temperature are aggravated by other factors, such as glycine infusion in transurethral resection, temperature can decrease even more. Preoperative warming prevents hypothermia, lowering the temperature gradient between core and peripheral compartments and reducing thermal redistribution. The most recent clinical practice guidelines advocate for active prewarming before induction of general anaesthesia since it is very effective in preventing perioperative hypothermia. However, the ideal warming time prior to the induction of anesthesia has long been investigated. This study aims to evaluate the optimal time period of preoperative forced-air warming to reduce the incidence of hypothermia at the end of surgery in patients submitted to transurethral resection. This is a clinical trial comparing different time periods of prewarming in patients submitted to undergo elective transurethral resection. We will compare different time periods: 0 minutes (control group), 15 minutes, 30 minutes and 45 minutes. 144 patients are going to be included in this study (36 patients in each group). Measurement of temperature will be performed using a tympanic thermometer. Patients will be followed throughout their hospital admission. Data will be recorded using a validated instrument and will be analysed using the statistics program R Core Team.

DETAILED DESCRIPTION:
Maintaining patient's temperature above 36 grades Celsius throughout the perioperative period is challenging. Thus, it is essential to monitor temperature in order to be able to take measures to avoid the appearance of hypothermia. Once the temperature has decreased, its treatment is difficult since the application of heat to the body surface takes a long time to reach the core thermal compartment. Intraoperative warming alone cannot avoid postoperative hypothermia. The application of forced-air warming system during the preoperative period has been shown to be the most effective measure to prevent hypothermia and maintain intraoperative normothermia. However, it would not be efficient to provide a long-time prewarming in short-term surgical procedures. Thus, the ideal warming time prior to the induction of anesthesia has long been investigated. Due to the searching of optimal prewarming time and the lack of evidence about the efficiency of prewarming in patients submitted to transurethral resection, the conductance of this clinical trial is justified.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective Transurethral resection under general or spinal anesthesia.
* Patients older tan 18 years old.
* American Society of Anesthesiologists physical status classification I - III.
* Absence of cognitive impairment.
* Written informed consent before enrollment.

Exclusion Criteria:

* American Society of Anesthesiologists physical status classification I - III.
* Pregnancy.
* Active infection.
* Intake of antipyretics within 24 hours before surgery.
* Neuropathy.
* Thyroid disorders.
* Peripheral vascular disease.
* Skin lesions.
* History of hypersensitivity to skin contact devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Differences in Body Temperature among different treatment groups (using tympanic and esophageal thermometers) | Throughout surgery, an average of 60 minutes.
  To assess the effects of prewarming in preventing drop of body temperature of patients undergoing elective transurethral resection.

SECONDARY OUTCOMES:
Length of stay in Post-Anesthetic Care Unit (in minutes) | Stay in Post-Anesthetic Care Unit, an average of 6 hours.
  To assess the effect of prewarming in the length of stay in the Post-Anesthetic Care Unit of patients undergoing elective transurethral resection.
Postoperative shivering (using a dichotomous scale: yes or no) | Immediate postoperative period, an average of 1 hour.
  To assess the effect of prewarming in the prevalence of postoperative shivering of patients undergoing elective transurethral resection.

CONTACTS AND LOCATIONS:
Overall Officials: Ángel Becerra, MD, Principal Investigator — Dr. Negrin University Hospital
Locations (1):
- Ángel Becerra, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data are to be shared with other researchers when required once the study is completed and global data are published.

REFERENCES:
- [Derived] Becerra A, Valencia L, Saavedra P, Rodriguez-Perez A, Villar J. Effect of prewarming on body temperature in short-term bladder or prostatic transurethral resection under general anesthesia: A randomized, double-blind, controlled trial. Sci Rep. 2021 Oct 21;11(1):20762. doi: 10.1038/s41598-021-00350-2. PMID 34675311